CLINICAL TRIAL: NCT06693674
Title: Effect of Sacubitril-Valsartan on Cardiac Structure and Function in Adults With Congenital Heart Disease
Brief Title: Effect of Sacubitril-Valsartan on Cardiac Structure and Function
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-009099; 5R01HL162830-02 (NIH)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Entresto (Experimental)
  Interventions: Drug: Entresto Pill
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Entresto Pill — Patients will take a 24/26 mg dose orally, twice daily, for weeks 1 and 2, 49/51 mg orally, twice daily, for weeks 3 and 4, and 97/103 mg orally twice daily, for the remaining 48 weeks (total duration: 52 weeks).
  Arms: Entresto
Other: Placebo — Patients taking placebo tablets will take 1 tablet orally, twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare changes in cardiac structure and function, biomarkers, and patient reported outcomes between adults with congenital heart disease (ACHD) randomized to angiotensin receptor-neprilysin inhibitor (ARNI) therapy vs placebo.

ELIGIBILITY:
Inclusion Criteria:

* Congenital Heart Disease Diagnosis
* Age 18 or Older

Exclusion Criteria:

* Stage IV chronic kidney disease defined as creatinine clearance <30 ml/min
* Hyperkalemia defined as serum potassium >5.2 mmol/l,
* Hypotension defined as systolic blood pressure <100 mmHg,
* History of angioedema related to previous ACE or ARB therapy
* Patients diagnosed with diabetes using Aliskiren,
* Pregnancy.
* Drug Therapies

  * Amifostine
  * Droperidol
  * Dantrolene
  * CYP3A4 Inhibitors
  * Obinutuzumab
  * Aliskiren
  * Lithium
  * Sparsentan
  * ACE inhibitor
  * ARB
  * ARNI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ventricular function | Baseline, Week 52
  Ventricular Function will be determined by indices of Right Ventricle (RV) and Left Ventricle (LV) systolic and diastolic function indices acquired from CMRI and transthoracic echocardiographic imaging.
Ventricular structure | Baseline, Week 52
  Ventricular structure will be determined by Right Ventricle (RV) and Left Ventricle (LV) size and wall thickness acquired from CMRI and transthoracic echocardiographic imaging.
Change from baseline in Hs-Troponin | Baseline, Week 52
  Hs-Troponin will be determined by blood specimen and will be measured in ng/L. A higher value indicates damage to the heart.
Change from baseline in Galectin 3 | Baseline, Week 52
  Galectin 3 will be determined by blood specimen and will be measure in ng/mL. A higher value indicates a higher severity of heart disease.
Change from baseline in Cystatin C | Baseline, Week 52
  Cystatin C will be determined by blood specimen and measured in mg/L. A lower value reflects better kidney function.
Change in baseline in Soluble ST-2 (sST-2) | Baseline, Week 52
  Soluble ST-2 (sST-2) will be determined by blood specimen and measured in ng/mL. A higher value indicates a higher severity of heart failure.
Patient reported outcomes | Baseline, Week 52
  Patient reported outcomes will be determined by a quality-of-life questionnaire. A self-assessment survey to assess the extent to which heart failure (HF) affects the patient's activities of daily living and quality of life. The questionnaire is 12 questions and a lower score reflects more severe the limitations on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No